CLINICAL TRIAL: NCT01627574
Title: Contraceptive Awareness and Reproductive Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Brown University (Other)
Responsible Party: Principal Investigator, Lynda Stein, Ph.D., Professor, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD065942; R01HD065942 (NIH)
Record Dates: First submitted 2012-06-15; First posted 2012-06-26 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy; Sexually Transmitted Infections
Keywords: Pregnancy; STI prevention; adolescents; probation
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Intervention (Experimental): There are two, 45-60 minute sessions of tailored Motivational Interviewing (MI). The first session occurs at the enrollment of the study, the second at 3 month follow-up.
  Interventions: Behavioral: Motivational Intervention
- Didactic Educational Intervention (Active Comparator): There are two, 45-60 minute sessions of didactic educational intervention related to promoting awareness for sexual health involving contraception and STI prevention. The first session occurs at the enrollment of the study, the second at 3 month follow-up.
  Interventions: Behavioral: Didactic Educational Intervention

INTERVENTIONS:
Behavioral: Motivational Intervention — There are two, 45-60 minutes sessions of tailored MI that occur at the enrollment of the study, and at 3 month follow-up.
  Other Names: Motivational Interviewing (MI)
  Arms: Motivational Intervention
Behavioral: Didactic Educational Intervention — There are two, 45-60 minute didactic sessions designed to provide information and awareness for sexual health involving contraception and STI prevention. The first session occurs after enrollment in the study, the second at 3 month follow-up.
  Other Names: Awareness of Sexual Health (ASH)
  Arms: Didactic Educational Intervention

SUMMARY:
The long-term objectives of this research are to develop effective treatments to reduce unplanned pregnancy and Sexually Transmitted Infections (STIs) for a highly under-served at-risk youth population.

DETAILED DESCRIPTION:
This trial will evaluate a Motivational Interviewing (MI) intervention designed to improve contraceptive use and decrease STIs for at-risk youth for both those who do and do not want a pregnancy. Those interested in becoming pregnant will be counseled in the risks associated with teen pregnancy and what it means to have a healthy pregnancy and raise a child. The investigators will utilize Title X programs in Rhode Island to provide reproductive health services in the community. The investigators will recruit 250 at risk youth from RI Juvenile Probation Department (JPD), RI group homes and alternative schools, Job Corps of Rhode Island, and Community Mental Health Centers and randomize them to two interventions: two sessions of personalized MI or two sessions of Awareness for Sexual Health (ASH), both delivered individually by trained counselors. MI is based on the principles of the Transtheoretical Model (TTM) and on MI, an empirically supported counseling technique designed to enhance readiness to change targeted behaviors. ASH provides didactic information about contraception, STI prevention and abstinence, and is intended to control for the effects of assessment and attention.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 14-21;
* 2) Currently sexually active with males defined as having had coital sex and intending to have coital sex within the next 6 months;
* 3) Willing to comply with protocol, follow-up assessments, and provide at least one locator; and
* 4) Fluent in English.

Exclusion Criteria:

* 1) Inability to give informed consent secondary to organic brain dysfunction, or active psychosis or otherwise not able to participate in the intervention or assessments (deaf, blind, or impaired communication skills that preclude participation in assessment or counseling);
* 2) Girls who are not sexually active; or
* 3) Currently pregnant.

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 272 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Stein, Ph.D., Principal Investigator — University of Rhode Island
Locations (5):
- United States (5):
  - Juvenile Probation, Cranston, Rhode Island
  - Exeter Job Corps, Exeter, Rhode Island
  - Family Services of Rhode Island (i.e. group homes), Providence, Rhode Island
  - MET Schools (i.e., network of alternative schools throughout Providence and Newport), Providence, Rhode Island
  - Community Care Alliance (i.e., Community Mental Health Center), Woonsocket, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delaney DJ, Stein LAR, Bassett SS, Clarke JG. Motivational interviewing for family planning and reducing risky sexual behavior among incarcerated men nearing release: A randomized controlled pilot study. Psychol Serv. 2023 Aug;20(3):538-552. doi: 10.1037/ser0000552. Epub 2021 Nov 4. PMID 34735198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This project enrolled 272 at-risk females aged 14-21. Participants were eligible if they had sexual intercourse with a male partner in the past four months, were not pregnant and intended to have intercourse with a male in the next 6 months. Recruitment began in February of 2013 and the last participant was recruited in August of 2017.
Period: Overall Study
Arm/Group | Motivational Intervention | Didactic Educational Intervention
Started | 142 | 130
Completed | 121 | 112
Not Completed | 21 | 18
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Lost to Follow-up | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Intervention | Didactic Educational Intervention | Total
Number analyzed (Participants) | 142 | 130 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.97 (1.71) | 16.99 (1.70) | 16.98 (1.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 130 | 272
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69 | 51 | 120
  Not Hispanic or Latino | 73 | 79 | 152
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 26 | 32 | 58
  White | 48 | 47 | 95
  More than one race | 52 | 40 | 92
  Unknown or Not Reported | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 142 | 130 | 272

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Continuous Use of Highly Effective Contraceptives Over 9 Months.
Description: Using the Timeline Followback (TLFB): Contraceptive use was measured via a calendar recall for both interventions.Continuous use of highly effective contraceptives at 9 Month follow up is determined if a participant remains on a highly effective contraceptive for 9 months. A participant switching from one highly effective contraceptive method to another is recorded as maintaining continuous contraceptive use at follow-up if she switches methods during times when the original method is still effective.
Time Frame: 9 month follow-up
Population: Continuous use of highly effective birth control is defined as those who are using effective birth control for 6 months or more. Thus this analysis only includes participants who initiated effective birth control for at least 6 months of data collection.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Intervention | Didactic Educational Intervention
Number analyzed (Participants) | 112 | 94
Participants | 39 | 29
Statistical Analysis 1: Comparison: Motivational Intervention vs Didactic Educational Intervention; Test type: Superiority; p > .05, Chi-squared, Corrected; Risk Ratio, log = .281, 95% CI 2-sided [.056 to 1.42], Standard Error of Mean .07

2. Primary Outcome: Number of Participants With a Positive STI Test After A Baseline Negative Test.
Description: Conducted STI testing for T. vaginalis, N. gonorrhoeae, and C. trachomatis through urine specimen collection. If a participant is diagnosed with an STI at baseline the youth will be referred for treatment at a Title X clinic and will be retested at the next follow-up visit. Any positive test after a baseline negative test will be documented as an incident infection.
Time Frame: 9 month follow-up
Population: Analysis conducted on all participants who provided a urine sample at baseline. 1 participant refused.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Intervention | Didactic Educational Intervention
Number analyzed (Participants) | 142 | 129
Participants | 18 | 13

3. Primary Outcome: Number of Participants Who Initiated a Highly Effective Contraceptive Post Treatment in 9 Months.
Description: Using the Timeline Followback (TLFB): The types of contraceptives used was captured via a calendar recall for both interventions. Initiation of highly effective contraceptives is determined if a participant ever endorses beginning a highly effective contraceptive at any time within 9 months.
Time Frame: 9 month follow up
Population: Analysis conducted on participants who initiated highly effective contraceptive use post treatment intervention. Those who initiated highly effective contraceptives at baseline (pre treatment) were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Intervention | Didactic Educational Intervention
Number analyzed (Participants) | 85 | 77
Participants | 61 | 51

4. Secondary Outcome: Number of Participants With a Positive Pregnancy Test After Baseline Assessment
Description: The secondary outcome is pregnancy as documented by a positive pregnancy test by at follow-up visit. Pregnancy tests were administered by urine collection and Home Pregnancy Test sticks.
Time Frame: 9 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Intervention | Didactic Educational Intervention
Number analyzed (Participants) | 142 | 130
Participants | 6 | 10

5. Secondary Outcome: Number of Participants Who Used Condoms 100% of the Time Thus Reducing the Risk of STIs.
Description: Using the Timeline Followback (TLFB): Condom use was measured via a calendar recall for both interventions. Participants indicate whether or not condoms were used each time sex was reported.
Time Frame: 9 month follow up
Reporting Status: Not Posted, anticipated posting 2025-11

6. Secondary Outcome: Number of Participants Who Reported Any Occasion of Substance Use and no Condom Use at the Time of Sex.
Description: Using the Timeline Follow-back (TLFB): Condom and substance use were measured via a calendar recall for both interventions. Participants indicate whether or not condoms and substances were used each time sex was reported.
Time Frame: 9 month follow-up
Reporting Status: Not Posted, anticipated posting 2025-11

ADVERSE EVENTS:
Time Frame: Clients were assessed over a 9 month period.
Arm/Group | Motivational Intervention | Didactic Educational Intervention
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/130
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/130
Other Adverse Events (participants affected / at risk) | 0/142 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT01627574/Prot_SAP_001.pdf